CLINICAL TRIAL: NCT05462613
Title: Induction Regorafenib in Combination With Metronomic Cyclophosphamide, Capecitabine, and Low-dose Aspirin Followed by Chemotherapy in Second Line Metastatic Colorectal Cancer Carcinoma An Open-label Randomized Phase II-III Study
Brief Title: Regorafenib With Low-dose Chemotherapies and Aspirin Followed by Standard Chemotherapies in Metastatic Colorectal Cancer
Acronym: REPROGRAM-02
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/702
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection; regorafenib; Aspirin; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Regorafenib + metronomic Capecitabine + metronomic Cyclophosphamide + low-dose Aspirin followed by second line of chemotherapy (Bevacizumab + FOLFOX or FOLFIRI)
  Interventions: Other: quality of life questionnaires; Procedure: Blood sample; Drug: Regorafenib; Drug: Metronomic chemotherapies; Drug: Aspirin; Drug: Bevacizumab; Drug: FOLFIRI or FOLFOX
- Control (Active Comparator): Second line of chemotherapy (Bevacizumab + FOLFOX or FOLFIRI)
  Interventions: Other: quality of life questionnaires; Procedure: Blood sample; Drug: Bevacizumab; Drug: FOLFIRI or FOLFOX

INTERVENTIONS:
Other: quality of life questionnaires — EORTC QLQ-C30 questionnaire (Quality of life questionnaire- Cancer 30) CR29 questionnaire (Colo-rectal cancer 29) EQ-5D3L questionnaire (EuroQol-5 Dimensions, 3 levels)
Procedure: Blood sample — Blood sample for plasma collection Blood sample for ctDNA (circulating tumoral DNA) collection
Drug: Regorafenib — - Regorafenib will be administered 3 weeks out of 4 for two months or unacceptable toxicity.
  * For the first cycle: regorafenib will be administered according to the "REDOS" schedule (80 mg daily for week 1, 120 mg daily for week 2 and 160 mg daily for the third week of the first cycle).
  * For the second cycle: regorafenib will be administered at 160mg in the absence of significant toxicity during cycle 1 or at a 80/120mg daily dose according to toxicity observed with the last dose used in the first cycle.
  Arms: Experimental
Drug: Metronomic chemotherapies — * Capecitabine: 625mg/m²/orally twice daily continuously during the first two months
  * Cyclophosphamide: 50 mg per os, daily, for two months
  Arms: Experimental
Drug: Aspirin — 75 mg orally and daily during two months
  Arms: Experimental
Drug: Bevacizumab — 5 mg/Kg every 2 weeks according to investigator practice, until disease progression or unacceptable toxicity
Drug: FOLFIRI or FOLFOX — every 2 weeks according to investigator practice

SUMMARY:
This study evaluates the interest of regorafenib in combination of metronomic chemotherapies and low-dose aspirin as a 2 months induction therapy before chemotherapy initiation in the second-line metastatic colorectal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven metastatic colorectal cancer in progression after a first line of chemotherapy +/- targeted therapy
2. Patients must have been treated for their metastatic disease with one of the following regimens as first-line therapy:

   * FOLFOX (Oxaliplatine, 5-Fluoro-uracil)
   * FOLFIRI (Irinotecan, 5-Fluoro-uracil)
   * FOLFIRINOX (Irinotecan, oxaplipatin, 5-Fluoro-uracil) or FOLFOXIRI (irinotecan, oxaliplatin, 5-Fluoro-uracil)
   * FOLFOX and anti-VEGFA (bevacizumab only)
   * FOLFIRI and anti-VEGFA (bevacizumab only)
   * FOLFIRINOX or FOLFOXIRI and anti-VEGFA (bevacizumab only)
   * FOLFOX and anti-EGFR (Epiderman Growth Factor Recepto)
   * FOLFIRI and anti-EGFR
   * FOLFIRINOX or FOLFOXIRI and anti-EGFR

   Of note, a chemotherapy prescribed for metastases occurring within six months after the end of an adjuvant chemotherapy are considered as a second line of therapy.
3. Patients should have a history of resistance to first line chemotherapy defined by:

   * Disease progression during the first line of their metastatic disease, less than 3 months after the last exposition to chemotherapy (even a chemotherapy regimen mentioned above or a 5-Fluoro-uracil-based maintenance therapy).
   * Disease relapse within 6 months after the end of an adjuvant FOLFOX based chemotherapy.
   * Disease relapse within 6 months after the surgical resection of metastases following a first line of chemotherapy.
4. Life expectancy of at least 3 months
5. Female or male with age ≥18 years old
6. Performance status Eastern Cooperative Oncology Group World Health Organization (ECOG-WHO) ≤1 (Appendix 1),
7. Measurable disease defined according to RECIST v1.1 (scanner or MRI)
8. Molecular status: patients eligible should have microsatellite-stable (MSS) status, absence of BRAF V600E (B(Raf gene, val600-to-glu) mutation and a known RAS (Retrovirus Associated Sequences) status.
9. Adequate bone marrow, liver and renal functions.

   * Haemoglobin ≥ 9 g/dL; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L
   * Total serum bilirubin ≤ 1.5 times upper normal value (ULN), serum alkaline phosphatase < 5 times ULN, aminotransferases (AST/ALT) ≤ 3 × ULN in absence of hepatic metastasis or ≤ 5 if presence of hepatic lesions
   * Cockcroft glomerular filtration rate > 50 ml/min
   * Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour
10. No contraindication to Iodine contrast media injection during CT
11. For female patients of childbearing potential, negative pregnancy test within 14 days before starting the study drug through at 210 days after the last dose of regorafenib. Men and women are required to use adequate birth control during the study (when applicable),
12. Signed and dated informed consent,
13. Ability to comply with the study protocol, in the Investigator's judgment.
14. Registration in a national health care system (CMU included).

Exclusion Criteria:

1. Diagnosis of additional malignancy within 2 years prior to the inclusion (exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical and/or bladder cancer),
2. Current participation in a study of an investigational agent. Patients might be included at least 21 days following the last investigational agent administration.
3. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial;
4. Patient under judicial protection (curators, autorship) and/or deprived of freedom,
5. Planned surgical procedure within the first month of treatment or any procedure that might change the timing of regorafenib administration during the first month of treatment,
6. Previous exposure to regorafenib,
7. Previous exposure to other anti-angiogenic treatment than bevacizumab,
8. Complete deficit in dihydropyrimidine dehydrogenase (DPD),
9. Major surgical procedure, open biopsy or significant traumatic injury within 28 days before start of study medication,
10. Pregnant or breast-feeding subjects,
11. Congestive Heart Failure ≥ New York Heart Association (NYHA) class 2, unstable angina (anginal symptomatology at rest),
12. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months),
13. Myocardial infarction less than 6 months before start of study drug,
14. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted),
15. Uncontrolled hypertension (Systolic blood pressure >150 mmHg and/or diastolic pressure >100 mmHg despite optimal medical management), or history of hypertensive crisis, or hypertensive encephalopathy
16. Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE grade 2 dyspnea),
17. Ongoing infection >grade 2 CTCAE V5 (Appendix 6 ),
18. Known History of human immunodeficiency virus (HIV) infection,
19. Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy,
20. Subjects with seizure disorder requiring medication,
21. History of organ allograft,
22. Subjects with evidence or history of any bleeding diathesis, irrespective of severity,
23. Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication,
24. Serious, Non-healing wound, active ulcer or untreated bone fracture,
25. History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to inclusion,
26. Dehydration CTCAE v4 grade ≥1,
27. Known hypersensitivity to any of the study drugs, study drug classes or excipient in the formulation,
28. Interstitial lung disease with ongoing signs or symptoms,
29. Persistent proteinuria of CTCAE Grade 3 (>3.5 g/24 hours),
30. Subject unable to swallow oral medications,
31. Any malabsorption condition, unresolved toxicity higher than CTCAE (V4) Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neuropathy ≤ Grade 2,
32. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 3 weeks,
33. Treatment with any other investigational medicinal product within 28 days prior to study entry, EXCEPT for ASPIRIN,
34. Co-administration of drugs potentially interacting with regorafenib i.e. CYP3A4 or UGT1A9 (UDP-glucuronosyltransferase 1-9) inducers/inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
best objective response during treatment period (phase II) | during treatment period (from first treatment administration and disease progression, an average of 14 months
  the best response rate evaluated with RECIST v1.1 criteria per an independent radiologist committee during the treatment period defined as the number of with complete response (CR) or partial response (PR) as best response divided by the total number of patients evaluable. Patients for whom best overall tumor response is not CR or PR will be considered non-responders.
overall survival (OS) (phase III) | through study completion, an average of 64 months
  Overall survival is defined as the time from the randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU de Besançon, Besançon
  - CHU Estain, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Nord Franche Comté, Montbéliard
  - CHU Montpellier, Montpellier
  - Groupe hospitalier de la région de Mulhouse et Sud Alsace, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital la Pitié-Salpétrière, Paris
  - Hôpital Saint antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Hôpital FOCH, Suresnes

IPD SHARING:
Plan to Share IPD: No